CLINICAL TRIAL: NCT05219929
Title: T4 - Tetracycline Treatment Tolerability Trial A Pilot Study Examining the Feasibility and Tolerability of Tetracycline Therapy in Post-Treatment Lyme Disease (PTLD)
Brief Title: Tetracycline Treatment Tolerability Trial
Acronym: T-4
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Steve and Alexandra Cohen Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: IRB00288079
Record Dates: First submitted 2022-01-21; First posted 2022-02-02 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Post-Treatment Lyme Disease
MeSH Terms: conditions — Post-Lyme Disease Syndrome | interventions — Tetracycline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tetracycline First (Active Comparator): Tetracycline for first 3 months, placebo for second 3 months.
  Interventions: Drug: Tetracycline 500 Mg; Other: Placebo
- Placebo First (Placebo Comparator): Placebo for first 3 months, tetracycline for second 3 months.
  Interventions: Drug: Tetracycline 500 Mg; Other: Placebo

INTERVENTIONS:
Drug: Tetracycline 500 Mg — 500 mg three times daily
Other: Placebo — Placebo for Tetracycline given same way as Tetracycline.

SUMMARY:
Randomized, double-blind, placebo-controlled study (with a one-week washout period) where subjects receive either 3 months of tetracycline or 3 months of placebo. After the 3 month primary endpoint, in the follow-up period, patients will be assigned to the alternate treatment for 3 months with blind maintained.

DETAILED DESCRIPTION:
There is precedent for the use of tetracycline class antibiotics as an anti-inflammatory agent in chronic illnesses including dermatologic and rheumatologic illnesses. The 2015 American College of Rheumatology Guideline for the Treatment of Rheumatoid Arthritis (RA) includes long-term therapy with tetracycline in its treatment recommendations. This class of antibiotics has known anti-inflammatory effect in addition to its antimicrobial properties. Tetracyclines, in particular minocycline, have been associated with a significant improvement in disease activity in RA with no increased risk of adverse effects.

To date, no clinical trials have examined the benefit of extended duration; i.e. >4 weeks tetracycline therapy in PTLD. Concerns over side effects and the development of antibiotic-resistance and superinfections such as Clostridioides difficile have limited the use of long-term antibiotics, including tetracycline. There is a large body of literature on tetracycline and other drugs in this class regarding the drugs' anti-inflammatory properties and potential benefit in several non-infectious diseases such cerebrovascular disease, rheumatoid arthritis, and rosacea.

The investigators believe that this deserves further study. Initially, the investigators propose this pilot study to examine the feasibility and tolerability of tetracycline treatment in PTLD Secondarily, the investigators propose to assess preliminary data on the efficacy of 3 months duration tetracycline treatment in reducing PTLD symptoms at (1) the end of the three-month treatment period, and (2) rate of change during the 1st 3 months of treatment.

Lastly, as an exploration, the investigators will explore in the follow-up period the return of symptoms after the completion of the 3 month tetracycline and the effect of 3 months of tetracycline in the placebo arm.

The investigators hypothesize that a tetracycline study over a 4 year interval will be feasible to conduct and tolerable to patients. Secondarily, the investigators hypothesize that 3 months of tetracycline treatment will be associated with greater improvements in fatigue, symptom burden and functional impact than placebo. This research is important because the long-term sequelae of LD are debilitating to patients and costly to society.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 to 80 years of age
* Meet criteria operationalized from the Infectious Diseases Society of America (IDSA) case definition for PTLD (ref) previously treated with at least one recommended course of antibiotic therapy.
* Have persistent symptoms in at least the last month. "Currently have at least one symptom attributed to Lyme disease that a) you've experienced in the past month and b) limits your daily functioning at least half the time when its present"
* Fatigue Severity Scale survey score of at least 4.0 signifying moderate or greater severity of fatigue.
* Medical Records documented history of definite or probable Lyme disease with onset starts in the last 5 years, with symptoms developing within 1 year of Lyme onset.

Definite LD. Medical record documented history of erythema migrans or medical record documented history of a Lyme disease compatible neurologic, cardiac or musculoskeletal manifestation of Lyme disease with a confirmatory 2-tier serology, modified 2-tier serologic test, or immunoglobulin G (IgG) western blot and a lack of alternative diagnosis Probable LD. Medical record documented history of Lyme disease with atypical or nonspecific manifestations with a confirmatory 2-tier serology, modified 2-tier serologic test, or IgG western blot and a lack of alternative diagnosis.

Exclusion Criteria:

* Medications:

No antibiotics in the prior 2 months No change in medications during the prior 4 months that might have an impact on primary and secondary outcome measures. See list. No immunosuppressive medications No medications that interact with tetracycline: atovaquone, retinoid medications taken by mouth (such as acitretin, isotretinoin), strontium, digoxin, kaolin pectin, warfarin Use of prescription or over the counter (OTC) medications containing calcium (i.e. Tums)

• History of the following conditions predating the diagnosis of Lyme disease: Myalgic encephalomyelitis/chronic fatigue syndrome Fibromyalgia Autoimmune disease

* Major psychiatric conditions Bipolar disorder, delusional disorder, schizophrenia Major depression Suicidal ideation with intent during the prior 6 months
* History of the following conditions in the last 4 months Alcohol or substance abuse Cancer (other than skin) Untreated HIV/AIDS Untreated moderate to severe sleep apnea Hepatitis A, B or C Pregnancy or intent to become pregnant Breastfeeding
* BMI greater than 40
* Other conditions at the discretion of the clinician

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-11-02 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Participant Retention | 36 months
  Number of participants retained.
Tolerability as assessed by number of side effects | 36 months
  Tolerability as assessed by number of side effects, as measured by Systematic Assessment for Treatment Emergent Events (SAFTEE).
Tolerability as assessed by severity of side effects | 36 months
  Tolerability as assessed by severity of side effects, as measured by SAFTEE.

SECONDARY OUTCOMES:
Fatigue as assessed by the Fatigue Severity Scale | 36 months
  A change of 0.7 in the Fatigue Severity Scale will be considered clinically significant

CONTACTS AND LOCATIONS:
Overall Officials: John N. Aucott, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Lyme Disease Research Center, Lutherville, Maryland, United States

IPD SHARING:
Plan to Share IPD: No